CLINICAL TRIAL: NCT06765369
Title: Predicting Microbiome-Associated Personalized Responses to the Mediterranean Diet
Brief Title: How the Mediterranean Diet Affects You: Predicting Responses Based on Your Microbiome
Acronym: MAP-Med
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Collaborators: University of Calgary (Other)
Responsible Party: Principal Investigator, Natasha Haskey, Research Associate, Department of Biology, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: H24-01007; POP23-11034 (Other Grant/Funding Number: Weston Family Foundation)
Record Dates: First submitted 2024-12-27; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: Healthy Individuals; Mediterranean diet; Westernized Diet; Predictive Microbiome
MeSH Terms: interventions — Diet, Mediterranean

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mediterranean Diet (Active Comparator): During the Mediterranean Diet (MD) phase, participants will receive three meals and two snacks per day for three weeks, adhering to the MD guidelines. To monitor compliance, participants will log their daily appetite and record any uneaten food. Additionally, participants will meet with the Research Coordinator weekly to receive guidance and support throughout the nutrition intervention.
  Interventions: Other: Mediterranean diet
- Westernized Diet (Active Comparator): During the Westernized Diet phase, participants will receive three meals and two snacks per day for three weeks, following a Westernized diet plan. To ensure compliance, participants will log their daily appetite and record any uneaten food. They will also meet with the Research Coordinator weekly for additional support and guidance.
  Interventions: Other: Westernized Diet
- Washout Period (No Intervention): This will be the period between two different interventions where participants will consume their usual diet while we wait for the participants' microbes to normalize after the first intervention before beginning the next one.

INTERVENTIONS:
Other: Mediterranean diet — The MD is characterized by increased consumption of legumes, whole grains, vegetables, fruits, nuts, seeds and olive oil, moderate consumption of fish, poultry and dairy foods, with low consumption of processed foods and red meat. The nutritional profile of the MD intervention will consist of 46% carbohydrates, 17% protein, and 35% fat. A significant focus on dietary fat consumption with maintaining an omega 6:3 ratio of approximately 3:1 or lower. The MD will provide fibre-rich foods to meet the fibre recommendations for Canadians (males: 30 grams/day, females: 21 grams/day)
  Arms: Mediterranean Diet
Other: Westernized Diet — The WD is characterized by increased consumption of highly processed foods, refined grains, red meats, processed meats, added sugars, added salt, high intake of omega-6 PUFA, accompanied by a reduction in fibre, fruits and vegetables, whole grains, fish, as well as nuts and seeds.The nutrition composition of the WD intervention will consist of 46% of calories derived from refined carbohydrates and added sugars, 17% protein (sourced from red and processed meats) and 35% fat. The fatty acid profile will be characterized by higher amounts of n-6 PUFAs while lacking in n-3 PUFAs and MUFAs, with a omega 6:3 ratio of 15-20:1.
  Arms: Westernized Diet

SUMMARY:
People respond differently to various diets-some may see significant benefits, while others may not. This project aims to personalize dietary recommendations by analyzing the gut microbiome to predict who will benefit most from the Mediterranean diet based on their unique biology, including their microbiome.

The study focuses on answering these key questions:

1. Are there specific microbes that influence who is most likely to benefit from the Mediterranean diet?
2. What changes occur in the gut microbiome when healthy individuals follow a Mediterranean diet?

To explore these questions, researchers will compare the effects of a Mediterranean diet to a Western-style diet. Participants will receive all their meals and snacks for the study to ensure accurate comparisons of how these diets impact the gut microbiome.

DETAILED DESCRIPTION:
Understanding the role of therapeutic dietary interventions in treating chronic diseases requires acknowledging that the response to nutrition varies in populations, subgroups and individual's. Varying responses to dietary intervention is dependent on interpersonal differences and environment. Personalized nutrition addresses these differences between individuals to maximize the benefits of dietary interventions. Many large, randomized controlled trials have effectively demonstrated that only 40% of a study cohort responds to dietary interventions, and lifestyle measures in regards to reducing disease risk. A more pragmatic approach to enhance the effectiveness of dietary treatment emerges by identifying microbiome-derived biomarkers capable of predicting and categorizing those most likely to benefit from specific nutritional interventions. Developing a predictive microbiome signature represents an advancement in this endeavour, offering the prospect of tailored, personalized nutrition interventions and a comprehensive understanding of the intricate interplay between diet, gut microbiota composition, and human health. Specifically, the Mediterranean diet (MD) has been investigated as a therapeutic diet for varying diseases due to its positive correlation with an array of health benefits. However, there is little consensus on specific microbial changes associated with the MD and how the MD alters the gut microbiome. This study aims to fill this knowledge gap that exists surrounding the MD and to determine a predictive microbiome associated with the MD. Ultimately producing a highly predictive microbiome signature that will have the ability to identifies those who will respond to the MD.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants, defined as free from cardiovascular disease, diabetes, and hypertension
* Body Mass Index of 20-25
* Between the ages 20-50 years
* Low adherence to the Mediterranean diet (MD serving score [MDSS] less than 10 points).
* Must live in the Okanagan area

Exclusion Criteria:

* Individuals with a self-reported history of irritable bowel syndrome, inflammatory bowel disease, Type-2 diabetes, kidney disease, intestinal obstruction, infectious gastroenteritis, colitis or gastritis, Clostridium difficile infection (recurrent) or Helicobacter pylori infection (untreated), malabsorption (such as celiac disease), major surgery of the GI tract, or colorectal cancer
* Oral antibiotics within three months of the intervention start date
* Individuals with any known food allergies, reported dietary intolerances of any kind, and those with eating disorders
* Pregnant or breastfeeding
* Participants with a high MDSS (> 10 points)
* Individuals who are intermittent fasting or refuse to follow the study protocol

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-01-08 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Microbiome - Microbial Diversity | Baseline, Week 3, Week 9 and Week 12
  Metagenomic sequencing will be employed to analyze stool samples, focusing on changes in the taxonomic composition of the gut microbiome in healthy individuals in response to interventions with the Mediterranean and Western diets.
Microbiome - Microbial Signature | Baseline, Week 3, Week 9 and Week 12
  Metagenomic sequencing will be utilized to analyze stool samples, aiming to identify microbial signatures of the gut microbiome in healthy individuals following interventions with the Mediterranean and Western diets.

SECONDARY OUTCOMES:
Metabolomics - Change in fecal metabolites | Baseline, Week 3, Week 9 and Week 12
  Fecal metabolites will be analyzed using a untargeted metabolomic platform with samples collected pre and post MD and Western diet. Quantification will be performed using untargeted reverse-phase ultrahigh-performance liquid chromatography tandem mass spectrometry (UHPLC-MS/MS).
Metabolomics - Change in serum metabolites | Baseline, Week 3, Week 9 and Week 12
  Serum metabolites will be analyzed using a untargeted metabolomic platform with samples collected pre and post MD and Western diet. Quantification will be performed using untargeted reverse-phase ultrahigh-performance liquid chromatography tandem mass spectrometry (UHPLC-MS/MS).
Change in Quality of Life | Baseline, Week 3, Week 9, Week 12
  Health-related quality of life will be measured using the 12-item short form-12 (SF-12). The SF-12 is comprised of two components: physical health and mental health. Scores range from 0 to 100, where a zero score indicates the lowest level of health and 100 indicates the highest level of health.
Dietary intake | Baseline, Week 9
  Dietary intake and supplement use will be evaluated at both baseline and week 9 using two non-consecutive 24-hour food recalls collected through the ASA-24 Canadian version. These assessments will establish participants' habitual dietary patterns and help monitor dietary consistency during the washout period.
Appetite rating | The Visual Analog Scales (VAS) for Appetite will be completed daily throughout the dietary intervention period, which includes 3 weeks on the Mediterranean diet and 3 weeks on the Western diet.
  Visual Analog Scales (VAS) for Appetite will be used to assess appetite of healthy participants in response to interventions with Mediterranean and Western diets. Higher values typically indicate greater intensity of the sensation being measured.
Change in Anxiety | Baseline, Week 3, Week 9 and Week 12
  Anxiety will be assessed by the GAD-7 (Generalized Anxiety Disorder-7). It is a self-reported screening tool used to measure the severity of generalized anxiety disorder (GAD) symptoms over the past two weeks. The total score ranges from 0 to 21. A score of 10 or higher typically indicates clinically significant anxiety and suggests the need for further evaluation or intervention..
Change in Depression | Baseline, Week 3, Week 9 and Week 12
  Depression levels will be assessed by PHQ-8 (Patient Health Questionnaire-8). It is a widely used self-report screening tool for assessing the severity of depressive symptoms over the past two weeks. The total score is the sum of all item responses, ranging from 0 to 24. A score of 10 or higher indicates the presence of clinically significant depressive symptoms and suggests the need for further evaluation or intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Natasha Haskey, RD PHD, Principal Investigator — University of British Columbia; Maitreyi Raman, MSc MD FRCPC, Principal Investigator — University of Calgary
Locations (1):
- University of British Columbia-Okanagan, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
All IPD used in the results of the publication will be shared
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From December 31, 2026 onward
Access Criteria: A proposal for planned analyses must be submitted to the PI's of this research.